CLINICAL TRIAL: NCT05196516
Title: Identification of Biomarkers for Post-COVID Conditions
Brief Title: Biomarkers for Post-COVID Conditions
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other); Skane University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SJ-947 (EMN-2021-07028)
Record Dates: First submitted 2022-01-14; First posted 2022-01-19 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: COVID-19; SARS-CoV-2; Biomarkers; Post-acute COVID-19 Syndrome
Keywords: Post-covid-19
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma and buffy coat are retained separately.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Individuals at age 18 to 65 with a SARS-CoV-2 infection proven by a polymerase chain reaction (PCR) test at least 12 weeks prior to inclusion and who have been referred to the clinic of post-COVID conditions.
- Controls: Healthy volunteers at age 18 to 65 with a SARS-CoV-2 infection proven by a PCR test at least 12 weeks prior to inclusion.

SUMMARY:
The COVID-19 infection affects humans differently. While some recover quickly and fully, others develop serious illnesses and late complications. The term late complications describe symptoms that last for 12 weeks or longer after COVID-19 infection is detected. The aim of the present project is to investigate whether it is possible to identify genetic factors that occur more frequently in people suffering from COVID-19 late complications than in those who do not develop late complications. The investigators aim to develop a genetic profile that identifies individuals at high risk for late complications of COVID-19. Number and nature of late complications will be analysed to identify patterns in the incidence of late complications associated with certain genetic traits. The study is designed as a case-control study and is expected to include 500 subjects between 18 and 65 years of age who at least 12 weeks ago tested positive for COVID-19; 250 who suffer from late complications and 250 who have fully recovered.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* SARS-CoV-2 infection proven by a PCR test at least 12 weeks prior to inclusion
* Only cases: Referred to the Clinic of post-COVID conditions located in Region Zealand, Denmark

Exclusion Criteria:

* Need of being on a respirator during infection with SARS-CoV-2
* Only controls: complain about long covid 12 weeks or more after proven infection with SARS-CoV-2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases are included from the population of patients referred to the Clinic of post-COVID conditions located in Region Zealand, Denmark.
  Controls are healthy volunteers included by a cohorte of 3500 individuals established by Department of Occupational and Environmental Health, Holbaek, Region Zealand.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Dyspnea | At inclusion
  Measured by means of Medical Research Council Dyspnoea Scale (MRC), which is a single-item, rated on a 5-point likert-scale in the range 1 to 5, with higher scores indicating worse symptoms.

SECONDARY OUTCOMES:
Hand grip strength (HGS) | At inclusion
  Measure the maximum isometric strength in the hand and forearm.
Psychic stress | At inclusion
  Measured by means of Kessler Psychological Distress Scale (K10), a 10-item questionnaire, scored on a 5-point Likert scale from 1 (None of the time) to 5 (All the time). The total score is in the range 10-50.
Cognitive impairment | At inclusion
  Measured by means of Montreal Cognitive Assessment (MOCA). The total score is in the range between zero and 30. A score of 26 and higher is considered normal.
Cognitive impairment | At inclusion
  Measured by means of Trail Making Test (TMT) which is scored by the number of seconds required to complete the task. Higher scores reveal greater impairment.
Cognitive impairment | At inclusion
  Measured by means of Symbol Digit Modalities Test (SDMT). The score is the correct number of substitutions in 90 s, and is in the range 0-110.
Physical and mental health | At inclusion
  Measured using the 12-point Short Form Health Survey (SF-12).
Ability to cope | At inclusion
  Measured by means of Coping Orientation to Problems Experienced Inventory (Brief COPE), a 28-items self-report questionnaire, scored on a 4-point Likert scale from 1 (I haven't been doing this at all) to 4 (I've been doing this a lot). The total score is in the range 28-112.
Level of Personality Functioning | At inclusion
  Measured by means of Level of Personality Functioning Scale - Brief Form (LPFS-BF), a 12-item self-report questionnaire, scored on a 4-point Likert scale from 1 (completely untrue) to 4 (completely true). The total score is in the range 12-48.
Work Rehabilitation | At inclusion
  Measured by means of Work Rehabilitation Questionnaire (WORQ).
Sexual function assessed by Female Sexel Function Index (FSFI_R) | At inclusion
  Measured by means of Female Sexel Function Index (FSFI_R) for women. FSFI-R is a 7-item self-report questionnaire, scored on a 5-point Likert scale from 1 to 5 .
Sexual function | At inclusion
  Measured by means of International Index of Erectile Function (IIEF-5) for men . IIEF-5 is a 5-item self-report questionnaire, scored on a 5-point Likert scale from 1 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Gesche Jürgens, Associate Professor, Ph.D., MD, Study Director — Clinical Pharmacology Unit, Zealand University Hospital, Roskilde, Denmark; Thomas Werge, Professor, Ph.D., Principal Investigator — Institute of Biological Psychiatry, Sct. Hans Hospital, Capital Region, Denmark; Fredrik Kahn, Associate Professor, Ph.D., MD, Principal Investigator — Department of infectious disease, Skåne University Hospital, Sweden
Locations (1):
- Zealand University Hospital, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
The investigators plan to make the results of the genetic analyzes available to other researchers as soon as the planned analyzes have been conducted.